CLINICAL TRIAL: NCT06948045
Title: Restructuring the Mandibular Angle in Facial Aging: a Novel Tecnique Using Poly-L-Lactic Acid
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Doris Hexsel (Other)
Collaborators: HEXSEL DERMATOLOGIC CLINICS RESEARCH DEPARTMENT (Unknown)
Responsible Party: Sponsor-Investigator, Doris Hexsel, Technical Director and Principal Investigator, Hexsel Dermatology Clinic
Organization: Hexsel Dermatology Clinic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08DPCHD2501
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Skin Laxity; Facial Aging
Keywords: Restructuring the mandibular angle in facial aging: a new technique using poly-L-lactic acid (PLLA); PLLA; poly-L-lactic acid; mandibular angle; facial aging
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Intervention group (Experimental): The 46 research participants, of both sexes, aged between 18 and 65 years, will be allocated to a single group in which all individuals will receive the study treatment sessions in the mandibular region with PLLA.
  Interventions: Procedure: PLLA application to the mandibular angle

INTERVENTIONS:
Procedure: PLLA application to the mandibular angle — The investigator will mark the application area by palpating the inferior and posterior boundaries of the face and the mandibular ramus, approximately 1 cm from these anatomical landmarks. The second PLLA injection point will be marked 1 cm from the inferior bony border of the mandible, anterior to the mandibular ligament. The demarcated area will be anesthetized with a local infiltration of 0.3-0.5 mL of 1% lidocaine with epinephrine, using a 30G needle. PLLA will then be reconstituted in 10 mL of sterile water for injection. Administration will be performed with a 30G needle inserted perpendicularly into the marked area until the supraperiosteal plane of the mandibular angle is reached, delivering a 0.7 mL bolus of the reconstituted product. At the second site-1 cm from the inferior bony border of the mandible, anterior to the mandibular ligament-a 0.2 mL dose of the reconstituted product will be injected.

SUMMARY:
Skin laxity is a common complaint among patients seeking aesthetic dermatological interventions, affecting the facial contour, especially in the mandibular angle, due to bone aging and the loss of tissue support in the lower third of the face. Facelift surgery is an effective method to address this issue, but it is invasive and may impact the definition of the jawline. As an alternative, poly-L-lactic acid (PLLA) stimulates collagen production, improving facial contour in a minimally invasive manner. This study aims to evaluate the safety and effectiveness of a new, low-cost, and quick application technique using poly-L-lactic acid in the mandibular angle and anterior to the mandibular ligament. The proposed technique seeks to enhance facial contour, provide an additional lifting effect, and contribute to overall facial rejuvenation. This is a clinical, prospective, and interventional study, allowing the analysis of clinical outcomes in terms of efficacy and safety. Twenty volunteers aged between 18 and 65, of both genders, with no restrictions on the use of collagen bio-stimulators, will be recruited. After confirming inclusion and exclusion criteria, participants will sign the Informed Consent Form (ICF) and be eligible for the study. The first intervention will occur at visit 2 (day 1), the second intervention at visit 3 (day 30 ± 15), and the third intervention will be performed as indicated at visit 4 (day 60 ± 15). Final follow-up will take place at visit 5 (day 90 ± 15). Questionnaires will be applied and photographs taken at all visits. Injections will be administered with poly-L-lactic acid in the mandibular angle region and anterior to the mandibular ligament. The study will be funded by the Research Department of the Hexsel Dermatology Clinic, and the data collected will be used to prepare an article for publication.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female individuals aged between 18 and 65 years of age.
2. Immunocompetent individuals.
3. Medical history and physical examination that, in the opinion of the investigator, do not prevent or contraindicate participation in the study or the use of the investigational product.
4. Female research participants of childbearing potential with a negative UPT at baseline (Day 1). These participants must use a highly effective contraceptive method throughout the study: combined oral contraceptives (estrogen and progesterone) or implanted/injectable contraceptives (with a stable dose for at least 1 month prior to study entry), bilateral tubal ligation, hormonal intrauterine device (inserted at least 1 month before entering the study), strict abstinence (at least 1 month prior to study entry and agreeing to continue throughout the study duration), vasectomized partner (at least 3 months before study entry), or condom use.
5. Women not of childbearing potential (e.g. postmenopausal with no menstrual bleeding for 1 year prior to study entry, hysterectomy, or bilateral oophorectomy).
6. Research participants who are willing and able to comply with the duration and procedures required by the study protocol.
7. Research participants who understand and sign the ICF and the ICF for image use authorization upon entering the study, before any investigational procedures are performed.

Exclusion Criteria:

1. Participants unable to understand the research protocol and/or follow the study schedule.
2. Pregnant or breastfeeding women, or those planning to become pregnant during the study period.
3. History of treatment in the past 6 months or planning to undergo procedures with lasers, intense pulsed light, radiofrequency, microfocused ultrasound, or deep chemical peels.
4. History of treatment with botulinum toxin on the face in the past 6 months or planning to undergo this procedure.
5. History of treatment with hyaluronic acid-based or other non-permanent dermal fillers on the face in the past 12 months, or planning to undergo this procedure.
6. History of treatment with collagen biostimulators on the face, such as poly-L-lactic acid (PLLA), calcium hydroxyapatite, or polycaprolactone, in the past 36 months, or planning to undergo this procedure.
7. History of treatment with or planning to use permanent fillers on the face.
8. Current use, use within the past 3 months, or planned use of collagen-based supplements.
9. Any surgical procedure or other treatment previously performed that has affected the area to be assessed in this study.
10. Active inflammation or infections in the facial region.
11. Severe psychiatric disorders.
12. Any other uncontrolled, chronic, or severe medical condition that, in the investigator's opinion, may interfere with the interpretation of the clinical study results or pose significant risk to the research participant.
13. History of sensitivity to any component of the product used in the study.
14. Vulnerable participants (such as those deprived of liberty), as defined in Section 1.61 of the International Conference on Harmonization (ICH) Guideline for Good Clinical Practice (GCP).
15. History of poor treatment adherence or demonstrated lack of cooperation in adhering to the study protocol.
16. Current participation in any other drug or device clinical study OR participation within 30 days prior to Day 1 or within an exclusion period of a previous clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of a new poly-L-lactic acid application technique through supraperiosteal injections along the contour of the mandibular angle and in the region anterior to the mandibular ligament. | 90 days
  To evaluate, through standardized comparative photographs before and after treatment sessions, using the Global Aesthetic Improvement Scale (GAIS).

SECONDARY OUTCOMES:
Assess patient satisfaction. Evaluate the safety of a new poly-L-lactic acid technique with supraperiosteal injections in the mandibular angle. Assess short-term outcomes after two or three intervention sessions based on clinical indications. | 90 days
  Assess the percentage of patients satisfied according to the study satisfaction questionnaire.
  Assess the overall frequency of adverse events related to the treatment and to the poly-L-lactic acid study product throughout the study period.
  Assess the percentage of patients demonstrating clinical improvement of at least 1 point in the final skin quality rating, based on an ordinal scale scored from 0 to 5.
  Assess the percentage of patients showing improvement in facial laxity using the Facial Laxity Grading Scale as assessed by the investigator.